CLINICAL TRIAL: NCT06002945
Title: Exploring Outcomes and Characteristics of Myasthenia Gravis 2
Acronym: EXPLORE-MG2
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Richard Nowak, Principal Investigator, Yale University
Other Study IDs: 2000026920; 1U54NS115054-01 (NIH)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Myasthenia Gravis
Keywords: Neuromuscular; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Muscle weakness; Autoimmune Diseases; Immune System Diseases
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Muscle Weakness; Autoimmune Diseases; Immune System Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurological Outpatients: Participants in this group will be recruited from the outpatient clinical population at MGNet participating sites. Treating physicians will make the initial determination of patients' potential eligibility to participate in the study.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Each blood draw will involve removing approximately 75 mL (5 tablespoons) of blood

SUMMARY:
The goal of this prospective observational study is to create a network repository of clinical data and biological samples to help researchers learn more about myasthenia gravis.

DETAILED DESCRIPTION:
The EXPLORE-MG2 (EXPLoring Outcomes and chaRactEristics of Myasthenia Gravis 2) study is a multi-center natural history study of myasthenia gravis (MG), a rare autoimmune disease characterized by weakness of the voluntary muscles. MG has a prevalence of approximately 14-40 per 100,000 people in the United States. There is no cure for MG, however, understanding the disease is crucial to pave the way for development of new therapies and a deeper mechanistic understanding to improve patient outcomes. Thus, EXPLORE-MG2 aims to accomplish comprehensive clinical phenotyping linked to bio-specimen collection in an effort to better understand disease characteristics and identify treatment predictive and responsive biomarkers. The primary purpose of this project is to create a network repository of data and biological samples to help researchers learn more about myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MG based on clinical presentation and seropositivity for MG associated autoantibodies (AChR binding, MuSK, or LRP4 antibodies), and/or a decremental response on repetitive nerve stimulation, positive single fiber electromyography (EMG) or positive edrophonium test. Signs and symptoms should not be better explained by another disease process.
* A) Diagnosed with MG within 2 years of study enrollment and with adequate records to document MG history (e.g., onset, MG meds) prior to enrollment at the discretion of the investigator.

or B) MuSK antibody, LRP4 antibody, or thymoma-associated MG at any point in the disease course. Patients with a diagnosis of MG more than 2 years prior to the first study visit who are expected to undergo a thymectomy may also be enrolled.

* Participant has the capacity to understand and sign a written informed consent form.
* Participant must be willing to complete the study and return for follow-up visits.

Exclusion Criteria:

* A history of chronic degenerative, psychiatric, or neurologic disorder other than MG that can produce weakness or fatigue that would confound outcome measure assessments or any disorder that interferes with participation in this protocol.
* Participant is unable or unwilling to comply with the study procedures.
* Treatment with any investigational agent within 4 weeks of the baseline visit or 5 half-lives of the investigational drug (whichever is longer).

  1. Participation in other observational studies is not exclusionary
  2. It is anticipated that some participants enrolled in EXPLORE-MG2 may be enrolled in future interventional trials while active in EXPLORE-MG2. This is acceptable. The exclusion only applies to starting EXPLORE-MG2 when participation in an interventional trial is imminent or active.
  3. If an EXPLORE-MG2 participant is later enrolled in an interventional trial, it will be at the investigator's discretion whether to continue collecting biosamples while the patient is participating in the interventional trial. Collection of natural history data should continue.
* Known active malignancy at enrollment other than skin cancer, low grade prostate cancer, or cervical cancer in situ. Thymoma is not included in this exclusion criteria.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates or that may affect the interpretation of the results or render the participant not an appropriate study participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be 18 years of age or older with a clinical diagnosis of a Myasthenia Gravis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The number of participants enrolled and serial blood reported at the conclusion of the enrollment period. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nowak, MD, Principal Investigator — Yale University; Vern Juel, MD, Principal Investigator — Duke University
Locations (10):
- United States (10):
  - University of California-Irvine, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No